CLINICAL TRIAL: NCT04199312
Title: Magnetic Muscle Stimulation of Abdominal Muscle
Acronym: MMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Discontinued due to business decision.
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA19-001
Record Dates: First submitted 2019-12-03; First posted 2019-12-13 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cohort 1: Magnetic Muscle Stimulation (MMS) (Experimental): Participants had a total of 4 MMS treatment sessions completed twice a week, within a 2-week period.
  Interventions: Device: Magnetic Muscle Stimulation (MMS) device
- Cohort 2: Magnetic Muscle Stimulation (MMS) (Experimental): Participants had 6 MMS treatment sessions completed twice a week, within a 3-week period.
  Interventions: Device: Magnetic Muscle Stimulation (MMS) device
- Cohort 3: Magnetic Muscle Stimulation (MMS) (Experimental): Participants had 8 MMS treatments completed twice per week within a 4-week period.
  Interventions: Device: Magnetic Muscle Stimulation (MMS) device

INTERVENTIONS:
Device: Magnetic Muscle Stimulation (MMS) device — The MMS device will be used to perform the treatments.

SUMMARY:
Evaluate the safety and efficacy of magnetic muscle stimulation (MMS) of abdominal muscle.

ELIGIBILITY:
Inclusion Criteria

* Male or female ≥ 22 years and ≤65 years of age.
* Subject has not had weight change exceeding 5% of body weight in the preceding month.
* Subject agrees to maintain body weight within 5% during the study by not making any changes in diet or exercise routine.
* Subject has a BMI ≤ 30 as determined at screening.
* Subject agrees to have photographs taken of the treatment area(s) during the scheduled time periods.
* Subject agrees to have MRI during the scheduled time periods.
* Subject agrees to refrain from any new abdominal muscle training exercises of the treatment area during the course of the study.
* Subject agrees to avoid sun tanning during the course of the study.
* Subject has read and signed the study written informed consent form.

Exclusion Criteria

* Subject has had a recent surgical procedure(s) in the area of intended treatment and muscle contractions may disrupt the healing process.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction procedure (e.g. CoolSculpting, SculpSure) in the area of intended treatment within the past 6 months.
* Subject needs to administer or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has had an intrauterine contraceptive device inserted or removed within the past month.
* Subject has a bleeding disorder or hemorrhagic condition
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has an active implanted electrical device such as a cardiac pacemaker, cochlear implant, intrathecal pump, hearing aids, defibrillator, or drug delivery system
* Subject has metal or electronic implants in or adjacent to the treatment area
* Subject has an abdominal hernia
* Subject has pulmonary insufficiency.
* Subject has a cardiac disorder.
* Subject has a malignant tumor.
* Subject has been diagnosed with a seizure disorder such as epilepsy.
* Subject currently has a fever.
* Subject is diagnosed with Grave's disease.
* Subject has a growth plate in the treatment area
* Subject is pregnant or intending to become pregnant during the study period (in the next 9 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject has any contraindications to MRI (e.g. metal implant, history of metal work or metal slivers in eye, prone to severe claustrophobia).
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any unapproved investigational device, investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Any other condition or laboratory value that would, in the professional opinion of the Investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Investigate MD, Scottsdale, Arizona
  - Innovation Research Center, Pleasanton, California
  - Laser and Skin Surgery Center of Northern California, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to 1 of 3 MMS treatment cohorts. As-Treated (Safety) Population includes all enrolled participants who received at least 1 treatment per protocol.
Groups:
- Cohort 1: Participants had 4 MMS treatment sessions completed twice a week, within a 2-week period.
- Cohort 2: Participants had 6 MMS treatment sessions completed twice a week, within a 3-week period.
- Cohort 3: Participants had 8 MMS treatments completed twice per week within a 4-week period.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 19 | 6 | 5
Completed | 19 | 6 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data presented here as planned and collected (all enrolled).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 19 | 6 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (11.3) | 43.5 (13.5) | 44.2 (14.2) | 45.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 4 | 3 | 25
  Male | 1 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 5 | 4 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Satisfaction Questionnaire From Baseline to 1-Month Post-Treatment Follow-up Visit
Description: Measurement of participant's perception about body shape, assessed using the Body Satisfaction Questionnaire (BSQ) at the 1-month post-treatment follow-up visit. The scale measures body image using a set of dichotomous items used to describe aspects of shape and appearance. The questionnaire has total score range from 10 to 50. An increase in score (when compared to baseline) reflects the participant's perceived improvement in appearance in the treated region (abdomen). Questionnaire results were tabulated as the numerical change between mean baseline scores and scores recorded at the 1-month post-treatment follow-up visit. A positive change reflects an increase in the body satisfaction questionnaire total score.
Time Frame: Baseline, 1-month post-treatment follow-up visit
Population: As-Treated Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 19 | 6 | 5
units on a scale | 6.2 (4.9) | 4.7 (6.1) | 2.8 (4.1)

2. Primary Outcome: Number of Participants With Device and/or Procedure Related Adverse Events (AEs) and Device-related Serious Adverse Events (SADEs)
Description: An AE was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, whether or not considered related to treatment. A serious adverse event (SAE) was an AE that resulted in death, serious deterioration in health, permanent impairment of a body structure/function, was life-threatening, required hospitalization or medical/surgical intervention, led to fetal distress or death, congenital abnormality, or birth defect. An ADE was any sign, symptom, or disease that was determined by the Investigator to have a causal relationship or possible causal relationship with the investigational device, including any AE resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the device or from use error or intentional misuse of the device. A SADE was an ADE that resulted in any of the consequences characteristic of an SAE.
Time Frame: AE information will be collected from the time of enrollment to the final follow-up visit at 3-months following the final treatment.
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 19 | 6 | 5
Participants
  Device and/ or Procedure Related AEs | 1 | 0 | 0
  SADEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of enrollment through the 8-week post-treatment follow-up visit, approximately 3 months.
Description: Safety data is presented here as planned and collected per protocol, by the total As-Treated Population (defined as all treated participants regardless of weight change).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/19 | 0/6 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=19) | Cohort 2 (N=6) | Cohort 3 (N=5)
Menstrual Cycle Irregularity (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT04199312/Prot_SAP_000.pdf